CLINICAL TRIAL: NCT03359590
Title: DPP-4 Inhibition With Sitagliptin and the Risk for Hypoglycaemia in the Fasting State in Subjects With Type 2 Diabetes Treated to Fasting Plasma Glucose Targets With Insulin Glargine and Metformin
Brief Title: Sitagliptin and the Risk for Hypoglycaemia in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DPP4-Hypo
Record Dates: First submitted 2017-11-24; First posted 2017-12-02 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Pharmacological Action
MeSH Terms: interventions — Sitagliptin Phosphate

STUDY DESIGN:
Intervention Model Description: This is a postmarketing phase 2 trial. The trial is designed as single centre, randomised, double blind, two-way treatment, placebo controlled crossover trial in subjects with type 2 diabetes mellitus treated to fasting plasma glucose targets with insulin glargine and metformin.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind randomised trial. Except for the unblinded persons involved in the preparation of the IMP (these persons are not involved in any other trial activities), everyone involved in the trial will be blinded until completion of the trial and the final data review.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin arm (Experimental): Sitagliptin 100 mg
  Interventions: Drug: Sitagliptin 100 mg
- Placebo arm (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin 100 mg — The treatment consists of sitagliptin tablets (100 mg/day) for up to 24 weeks.
  Arms: Sitagliptin arm
Drug: Placebo — The treatment consists of placebo tablets for up to 24 weeks.
  Arms: Placebo arm

SUMMARY:
Sitagliptin, through its effects on sensitizing alpha-cell sensitivity to glucose, can initiate counter-regulatory glucagon responses at higher glycemic thresholds, thus reducing the number of clinically apparent hypoglycemic episodes, and/or ameliorating the severity of hypoglycemic episodes in the case that they should occur. The endpoints have defined such that consequences of this hypothesis can be measured.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject with diabetes mellitus type 2.
* Age between 18 and 64 years, both inclusive.
* HbA1c <= 8.5%.
* Stable treatment with insulin glargine (any dose) and metformin (>= 1500 mg/day or at highest tolerated dose) for at least 3 months prior to inclusion into the trial with or without additional oral glucose-lowering agents (except thiazolidinediones).
* Considered generally healthy (apart from diabetes mellitus type 2 and associated conditions such as hypertension, hyperlipidaemia and hyperuricaemia) upon completion of medical history, physical examination, vital signs, ECG and analysis of laboratory safety variables, as judged by the Investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to sitagliptin or related products.
* More than one episode of severe hypoglycaemia with seizure, coma or requiring medical assistance of another person during the past 6 months or hypoglycaemic unawareness as judged by the Investigator.
* Current or previous treatment (less than 3 months prior to screening) with insulin products other than insulin glargine and/or with Glucagon-like peptide (GLP) 1 receptor agonists and/or with thiazolidinediones.
* Unwillingness to wash-off any oral glucose-lowering agents other than metformin.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kapitza, MD, Principal Investigator — Profil GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by use of the site specific database
Pre-assignment Details: All subjects underwent outpatient insulin titration during each treatment period. The aim was to find the insulin dose that, under these conditions, stabilised individual fasting plasma glucose for at least one week
Groups:
- Sequence 1: First intervention: treatment with sitagliptin tablets (100 mg/day) for up to 24 weeks.
  Washout 4 weeks Second intervention: treatment with placebo tablets for up to 24 weeks.
- Sequence 2: First intervention: treatment with placebo tablets for up to 24 weeks. Washout 4 weeks Second intervention: treatment with sitagliptin tablets (100 mg/day) for up to 24 weeks.
Period: First Intervention
Arm/Group | Sequence 1 | Sequence 2
Started | 10 | 10
Exposed | 9 | 10
Discontinued | 1 | 2
Completed | 9 | 8
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1
Period: Second Intervention
Arm/Group | Sequence 1 | Sequence 2
Started | 9 | 8
Exposed | 9 | 8
Discontinued | 0 | 0
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants of both arms are included here
Groups:
- All Study Participants: Drug: Sitagliptin or placebo
  The treatment consists of sitagliptin 100 mg/day or placebo for up to 24 weeks.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 20
Body mass index (BMI, kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 29.19 (4.139)
Waist circumference (cm) [Mean (Standard Deviation); unit: cm] | 105.9 (9.02)
Height (cm) [Mean (Standard Deviation); unit: cm] | 178.1 (9.20)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 92.32 (13.79)
HbA1c (%) [Mean (Standard Deviation); unit: percent] | 7.35 (0.661)

OUTCOME MEASURES:

1. Primary Outcome: The Frequency of Hypoglycaemic Episodes With Sitagliptin vs Placebo Treatment.
Description: The purpose of the trial was to test the influence of DPP-4 inhibition on the risk to develop hypoglycaemia. Chemical hypoglycaemic episodes (characterised by a plasma glucose nadir ≤70 mg/dL) occurring during the in-house periods of the subjects were compared.
Time Frame: during the two in-house periods (54 hs each) after treatment with sitagliptin or placebo for up to 24 weeks
Population: The per protocol analysis set comprised all subjects completing the trial.
Measure: Mean (Standard Deviation); unit: Hypoglycaemic episodes
Groups:
- Sitagliptin Arm: Drug: Sitagliptin
  The treatment consists of sitagliptin 100 mg/day up to a maximum of 24 weeks.
- Placebo Arm: Drug: Placebo
  The treatment consists of placebo up to a maximum of 24 weeks.
Arm/Group | Sitagliptin Arm | Placebo Arm
Number analyzed (Participants) | 17 | 18
Hypoglycaemic episodes | 5.35 (4.137) | 5.72 (3.045)

ADVERSE EVENTS:
Time Frame: For each participant from baseline to end of trial, with a range from 7-53 weeks per participant, on average 11 weeks
Description: In this report, only treatment-emergent adverse events (TEAEs) are reported, occurring after randomisation. No AEs were reported for the washout period.
Arm/Group | Sitagliptin Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/19
Other Adverse Events (participants affected / at risk) | 12/17 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin Arm (N=17) | Placebo Arm (N=19)
Coronary heart diesease (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin Arm (N=17) | Placebo Arm (N=19)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Decapitation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion site thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle contractions involuntary (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Allodynia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (4)
Headache (Nervous system disorders) | 6 (6) | 3 (3)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthostatic intolerance (Vascular disorders) | 1 (1) | 0 (0)
Syncope (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT03359590/Prot_SAP_000.pdf